CLINICAL TRIAL: NCT06131554
Title: A Multicenter, Randomized, Double-blinded, Positive-controlled Phase Ⅲ Clinical Trial to Evaluate Lot-to-lot Consistency, Immunogenicity and Safety of Group ACYW135 Meningococcal Conjugate Vaccine (CRM197) in Adults Aged 18 to 55 Years
Brief Title: A Clinical Trial to Evaluate the Immunogenicity and Safety of Group ACYW135 Meningococcal Conjugate Vaccine (CRM197) in Adults Aged 18 to 55 Years
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CanSino Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CTP-MCVF-006
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-08

CONDITIONS: Meningococcal Meningitis
Keywords: Vaccine; Positive controlled; Immunogenicity; Safety; 18-55 years
MeSH Terms: conditions — Meningitis, Meningococcal | interventions — CRM197 (non-toxic variant of diphtheria toxin); Meningococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- batch 1 of MCV4 (Experimental): 1 dose of Menhycia on Day 0
  Interventions: Biological: batch 1 of Group ACYW135 Meningococcal Conjugate Vaccine (CRM197) (MCV4)
- batch 2 of MCV4 (Experimental): 1 dose of Menhycia on Day 0
  Interventions: Biological: batch 2 of MCV4
- batch 3 of MCV4 (Experimental): 1 dose of Menhycia on Day 0
  Interventions: Biological: batch 3 of MCV4
- Meningococcal (Groups A, C, Y, and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine (Active Comparator): 1 dose of Menactra on Day 0
  Interventions: Biological: Meningococcal (Groups A, C, Y, and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine

INTERVENTIONS:
Biological: batch 1 of Group ACYW135 Meningococcal Conjugate Vaccine (CRM197) (MCV4) — 1 dose of Menhycia (0.5ml) on Day 0, Intramuscular injection
  Other Names: Menhycia
  Arms: batch 1 of MCV4
Biological: batch 2 of MCV4 — 1 dose of Menhycia (0.5ml) on Day 0, Intramuscular injection
  Other Names: Menhycia
  Arms: batch 2 of MCV4
Biological: batch 3 of MCV4 — 1 dose of Menhycia (0.5ml) on Day 0, Intramuscular injection
  Other Names: Menhycia
  Arms: batch 3 of MCV4
Biological: Meningococcal (Groups A, C, Y, and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine — 1 dose of Menactra (0.5ml) on Day 0, Intramuscular injection
  Other Names: Menactra
  Arms: Meningococcal (Groups A, C, Y, and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine

SUMMARY:
This is a multicenter, randomized, double-blinded, positive controlled study to evaluate the lot-to-lot consistency, immunogenicity and safety of Group ACYW135 Meningococcal Conjugate Vaccine (CRM197) in adults aged 18 to 55 years. Subjects will be randomized to receive investigational Lot 1, Lot 2, Lot 3 vaccine or control vaccine in a 1:1:1:1 ratio, with the subjects in experimental group randomly and equally assigned to three different batches of MCV4 for single-dose vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18-55 years old at the time of screening, who are in good health condition as determined by the study clinician.
* Participants who have not been vaccinated with any meningococcal vaccines (including but not limited to meningococcal group A and C conjugate vaccine, meningococcal group A and C polysaccharide vaccine, Group ACYW135 Meningococcal polysaccharide/conjugate vaccine).
* The participant or participant's legal guardian signs the informed consent form (ICF) and participant agrees to comply with the requirements of protocol and finish the 1-year follow-up.
* Participants who are willing to discuss medical history with investigators or doctors and allow access to all medical records relevant to this trial.
* Participants with child-bearing potential who are willing to practice adequate contraception methods from signing the ICF to 12 months after vaccination. This includes:

  1. Abstinence from penile-vaginal intercourse,
  2. Hormonal contraceptives such as oral contraceptives (the pill), injectables, implants, patches or estrogen vaginal ring (a ring-shaped hormonal contraceptive device that is used inside the vagina),
  3. Intrauterine device (IUD/Spiral),
  4. Male partner sterilization (vasectomy) prior to the female subject's entry into the study, and this male is the sole partner for that subject,
  5. Male condom combined with a vaginal spermicide (a substance that can kill the sperm cells inside the vagina) or female diaphragm, whether with or without a vaginal spermicide .
* Be able to communicate well with the investigator, and to understand and comply with the requirements of this clinical trial.

Exclusion Criteria:

* Axillary temperature >37.5°C (99°F).
* Have congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.
* A history of epilepsy, convulsions or history/family history of mental illness.
* Have meningitis or a history of meningitis illness.
* Positive result of urine pregnancy test (also required for women within one year of menopause), lactating women, or participant /his partner is planning to become pregnant within 1 year.
* Hypersensitivity to a component or excipient of the vaccine used in this clinical trial (mainly: group A, C, Y or W135 meningococcal capsular polysaccharide, diphtheria toxoid or diphtheria antigen, sucrose, mannitol, sodium chloride, dipotassium hydrogen phosphate trihydrate, potassium dihydrogen phosphate).
* In the past 6 months (internal time < 6 months), participants have received immunosuppressive treatment, cytotoxic treatment, glucocorticoid treatment, etc. (excluding local treatment, surface treatment of acute non-concurrent dermatitis, spray treatment of allergic rhinitis).
* Received or plan to receive blood/plasma products or immunoglobulins throughout the study period or 60 days prior to study vaccination.
* Use of non-prescription drugs such as antipyretic (e.g., acetaminophen) and anti-inflammatory drugs (e.g., ibuprofen, naproxen etc.) within 12 hours before the administration of vaccine.
* Have severe hypertension that is not controlled by medication (at the time of field measurement: systolic blood pressure ≥ 160 mmHg and diastolic blood pressure ≥ 100 mmHg).
* Suffering from a severe chronic disease or a condition that is in a progressive stage and cannot be well controlled, such as thyroid disease
* Participants with known or suspected diseases that are judged by the investigator to affect the vaccination assessment, for example, acute infectious diseases, severe respiratory disease, severe cardiovascular disease, severe allergic skin disease etc.
* History of serious adverse reactions associated with the vaccine and/or history of severe allergic reactions (e.g., systemic allergic reactions) to any component of the study vaccine.
* Immunocompromised individuals with known or suspected immunodeficiency as determined by medical history and/or physical examination (e.g., HIV infection, history of pancreatic, liver, spleen, kidney disease or history of resection).
* Positive for HIV, Hepatitis B, Hepatitis C or Syphilis.
* Bleeding constitution or condition associated with prolonged bleeding for which intramuscular injection is contraindicated in the opinion of the investigator.
* Administration of live attenuated vaccine within 14 days or other vaccines within 7 days.
* Participation in other studies involving interventional studies within 28 days prior to screening and/or during study participation.
* According to the judgment of the investigator, participants could be excluded due to various medical, psychological, social or other conditions that are contrary to the trial protocol or that affect the subject's ability to sign informed consent.
* Investigator site staff directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members，sponsor staff and their respective family members.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1480 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The geometric mean titer (GMT) of serogroup A, C, Y and W135 meningococcal rSBA titer in all participants. | Day 30 post vaccination
The seroconversion rate of serogroup A, C, Y, and W135 meningococcal rSBA titer. | Day 30 post vaccination
The incidence of adverse reactions (ARs) in all participants. | Within 7 days post vaccination

SECONDARY OUTCOMES:
The geometric mean fold increase (GMI) of serogroup A, C, Y and W135 meningococcal rSBA titer in all participants. | Day 30 post vaccination
The proportion of GMT ≥ 1:128 of serogroup A, C, Y and W135 meningococcal rSBA titer on day 30 post vaccination in all participants. | Day 30 post vaccination
The incidence of ARs and adverse events (AEs) in all participants. | Within 30 days post vaccination
The incidence of ARs in all participants. | Within 30 min post vaccination
The incidence of serious adverse events (SAEs) in all participants. | Within 365 days post vaccination
The GMT of serogroup A, C, Y and W135 meningococcal antibodies in the 480 subjects (120 of each subgroup,Immunopersistence group) | Day 90, day 180 and day 365 post vaccination
The GMI of serogroup A, C, Y and W135 meningococcal antibodies in the 480 subjects (120 of each subgroup,Immunopersistence group). | Day 90, day 180 and day 365 post vaccination
The proportion of GMT ≥ 1:128 of serogroup A, C, Y and W135 meningococcal antibodies in the 480 subjects (120 of each subgroup,Immunopersistence group). | Day 90, day 180 and day 365 post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Isti Suharjanti, Dr, Principal Investigator — Husada Utama Hospital
Locations (1):
- Husada Utama Hospital, Surabaya, Indonesia